CLINICAL TRIAL: NCT05800613
Title: Management of Ovarian Masses in Pediatric Patients: an Italian Survey
Acronym: OvaMa-PEDs
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Moro Francesca, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5003
Record Dates: First submitted 2023-03-24; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cysts; Pediatric ALL; Diagnosis
Keywords: ovarian cysts; Pediatric patients; Ultrasound; Survey
MeSH Terms: conditions — Ovarian Cysts; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Questionnaire

SUMMARY:
Objectives: The International Ovarian Tumor Analysis (IOTA) provides a specific terminology for adult ovarian masses, while, currently, there is no systematic classification for preoperative assessment of adnexal lesions in childhood and adolescence. This study aims to survey Italian pediatric surgeons to evaluate ovarian masses' management (from diagnosis to treatment) in patients aged 1-18.

Methods: A 27-question survey was distributed. It consisted of questions regarding the management and use of ultrasound and IOTA terminology in diagnosing ovarian masses in childhood and adolescence, in emergency regimes and in planned surgeries.

DETAILED DESCRIPTION:
PURPOSE AND OBJECTIVES OF THE CLINICAL TRIAL The aim of the present study is to propose a survey among Italian Pediatric Surgeons (inside the Società Italiana di Chirurgia Pediatrica-SICP) to evaluate the current management of ovarian masses in patients aged 1 -18, in terms of preoperative work up and surgical modalities.

EXPERIMENTAL DESIGN

PRIMARY OBJECTIVE:

To evaluate the current management of ovarian masses in patients aged between 1 and 18.

EXPERIMENTAL PLAN:

Observational study, survey.

SETTING:

This is an online survey designed using REDCap forms feature. Data will be collected in a period of 6 months. The informed consent forms for participation, use of personal data and the link for the questionnaire will be sent by e-mail to all Italian Pediatric Surgeons belonging to the SICP. The surgeons who accept to participate, will return both signed consent forms and a copy of their Identity Card.

The survey is divided into seven sections.

* Section 1: demographic data.
* Section 2: data on surgical background of the institution and the pediatric surgeons.
* Section 3: management of pediatric patients in emergency.
* Section 4: management of pediatric patients who had planned surgery.
* Section 5: additional management data.
* Section 6: knowledge of the IOTA group and terminology.
* Section 7: availability to participate in a multi-center retrospective study.

Questions asked for responses using yes/no, multiple-choice, or short freeform written answers. More than one response could be given for many questions, it is specified.

(The detailed description is reported in the attachment 1).

ELIGIBILITY:
Inclusion Criteria:

Pediatric surgeons who work in public hospitals that have managed or collaborated in the management of pediatric patients affected by ovarian cyst.

Signed informed consent for participation in the study and for the use of personal data.

Exclusion Criteria No answer and/or non-completion of the questionnaire within 1 month after sending our e-mail.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric surgeons who work in public hospitals that have managed or collaborated in the management of pediatric patients affected by ovarian cyst.
  Signed informed consent for participation in the study and for the use of personal data.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the current management of ovarian masses in patients aged between 1 and 18 | 6 months
  Collect data from the survey

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli, IRCCS, Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No